CLINICAL TRIAL: NCT05761275
Title: Assessment of Women's Sexual Quality of Life After Benign Adnexal Surgery Using vNOTES Approach in Comparison to Conventional Laparoscopy: a Randomized Controlled Trial
Brief Title: Assessment of Women's Sexual Quality of Life After Benign Adnexal Surgery Using vNOTES Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Dubuisson (Other)
Responsible Party: Sponsor-Investigator, Jean Dubuisson, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00407
Record Dates: First submitted 2023-01-10; First posted 2023-03-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic Disease; Adnexal Mass; Adnexal Cyst; Sexuality; Adnexal Diseases; Sexual Dysfunction; Quality of Life; Pathology; Dyspareunia; Pelvic Pain; Complication
MeSH Terms: conditions — Genital Diseases, Female; Sexuality; Adnexal Diseases; Sexual Dysfunction, Physiological; Dyspareunia; Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Abdominal Laparoscopy (Active Comparator): Use of conventional transabdominal laparoscopy as the surgical approach to perform the indicated procedure in the included patient with benign adnexal pathology (elective cystectomy/oophorectomy elective salpingectomy or tubal sterilization).
  Interventions: Procedure: Elective cystectomy; Procedure: Elective oophorectomy; Procedure: Elective salpingectomy; Procedure: Elective tubal sterilization
- vNOTES (Experimental): Use of vNOTES (Transvaginal Natural Orifice Transluminal Endoscopic Surgery) as the surgical approach to perform the indicated procedure in the included patient with benign adnexal pathology (elective cystectomy/oophorectomy elective salpingectomy or tubal sterilization).
  Interventions: Procedure: Elective cystectomy; Procedure: Elective oophorectomy; Procedure: Elective salpingectomy; Procedure: Elective tubal sterilization

INTERVENTIONS:
Procedure: Elective cystectomy — Adnexal cyst removal for presumed benign adnexal pathology.
Procedure: Elective oophorectomy — Ovarian removal for presumed benign adnexal pathology.
Procedure: Elective salpingectomy — Tubal removal for presumed benign adnexal pathology.
Procedure: Elective tubal sterilization — Tubal obstruction as a definitive contraceptive method (tubal cauterization with or without sectioning, partial or total removal of both tubes, or obstruction with small clips/ligatures).

SUMMARY:
Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is a recent innovation in minimally invasive surgery which has already proven its non-inferiority to conventional abdominal laparoscopy (CAL) for hysterectomy in terms of efficiency and safety. However, the investigators note a lack of medical literature and no specific randomized controlled trial (RCT) assessing women's sexual function after vNOTES for benign adnexal surgery.

The aim of this RCT is to confirm the non-inferiority of the vNOTES approach for benign adnexal pathology compared to CAL on women's sexual function. Secondary outcomes will evaluate vNOTES's efficiency, morbidity and postoperative complications compared to CAL for benign adnexal surgery. The relationship between adnexal mass morcellation/aspiration and the quality of the histological analysis on surgical specimens will also be evaluated as secondary outcome.

DETAILED DESCRIPTION:
This study focuses on women aged 18 to 70 who require surgery for benign adnexal disease (removal of an ovarian cyst, ovary and/or fallopian tube). This is a randomised study, i.e. each woman will be randomly assigned the surgical technique used for the planned operation, either vNOTES or conventional transabdominal laparoscopy.

Currently, there are no randomised clinical trials specifically investigating the impact on women's sexual quality of life after benign adnexal surgery compared to conventional transabdominal laparoscopy. Patients appear to be more reticent about the vaginal approach to surgery due to fear of possible alteration of their sexual activity afterwards. Indeed, their fears relate to the vaginal scarring that occurs during the vNOTES surgery. The vaginal scar could cause vaginal pain and pain during sexual intercourse, especially if there is a post-operative complication with the vaginal scar. The vaginal scar could also alter women's perception of their bodies during sexual intercourse. This study is necessary to answer these questions and increase women's acceptance of the vNOTES technique for benign adnexal surgery. In this way, women would benefit from the advantages of vNOTES without fearing an impact on their sexual quality of life.

The primary objective of this study is to demonstrate that the vNOTES technique, although using the vagina as an entry route, does not significantly alter the quality of sexual life of women after benign adnexal surgery compared to conventional transabdominal laparoscopy.

The secondary objectives of this study evaluate the effectiveness of vNOTES (impact on pain, length of stay after surgery and patient satisfaction), complications ( during surgery and up to 30 days after surgery), as well as the relationship between the need to cut the surgical specimen for extraction and the difficulty of microscopic analysis.

All participants in the study, regardless of the surgical technique assigned to them, will complete questionnaires to assess their quality of sexual life before surgery and at 3 and 6 months after surgery. These are the FSFI (female sexual function), CSI-16 (couple satisfaction) and a self-created questionnaire on pain during sex (dyspareunia). These questionnaires will determine whether there is a difference in the women's quality of sexual life before and after surgery, as well as comparing the two surgical techniques. The participants' general and medical data will be collected at the time of study enrolment, during hospitalisation and at one month after surgery to assess the secondary objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 70 years
* Discernment capacity with oral and written consent signed
* Heterosexual intercourse (with vaginal penetration) within four weeks prior to inclusion in the study

Exclusion Criteria:

* History of rectal surgery.
* Suspected rectovaginal/retrocervical endometriosis.
* History of brachytherapy or pelvic radiation.
* Suspected malignancy.
* History of severe pelvic inflammatory disease.
* Active lower genital tract infection.
* Pregnancy.
* Women who do not speak fluent French or English.
* Patients under tutelage (with or without capacity of judgement).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Women's quality of sexual life evaluation - Female Sexual Function Index (FSFI) | Preoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Female Sexual Function Index (FSFI) questionnaire.
  FSFI, created in 2000 by Raymond Rosen, is a reliable and complete multidimensional self-reported instrument for the measurement of female sexual function. It is validated in English and assesses 19 items divided into six domains of sexual function: (a) desire (2 items), (b) subjective arousal (4 items), (c) lubrication (4 items), (d) orgasm (3 items), (e) satisfaction (3 items) and (f) pain/discomfort (3 items). Each item focuses on the situation during the last 4 weeks. The total score is the sum of answers provided for each of the 6 domains. Lower is the score, worse is the patient's sexual function. A total score below 26 defines impaired sexual function.
Women's quality of sexual life evaluation - Female Sexual Function Index (FSFI) | 3 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Female Sexual Function Index (FSFI) questionnaire.
  FSFI, created in 2000 by Raymond Rosen, is a reliable and complete multidimensional self-reported instrument for the measurement of female sexual function. It is validated in English and assesses 19 items divided into six domains of sexual function: (a) desire (2 items), (b) subjective arousal (4 items), (c) lubrication (4 items), (d) orgasm (3 items), (e) satisfaction (3 items) and (f) pain/discomfort (3 items). Each item focuses on the situation during the last 4 weeks. The total score is the sum of answers provided for each of the 6 domains. Lower is the score, worse is the patient's sexual function. A total score below 26 defines impaired sexual function.
Women's quality of sexual life evaluation - Female Sexual Function Index (FSFI) | 6 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Female Sexual Function Index (FSFI) questionnaire.
  FSFI, created in 2000 by Raymond Rosen, is a reliable and complete multidimensional self-reported instrument for the measurement of female sexual function. It is validated in English and assesses 19 items divided into six domains of sexual function: (a) desire (2 items), (b) subjective arousal (4 items), (c) lubrication (4 items), (d) orgasm (3 items), (e) satisfaction (3 items) and (f) pain/discomfort (3 items). Each item focuses on the situation during the last 4 weeks. The total score is the sum of answers provided for each of the 6 domains. Lower is the score, worse is the patient's sexual function. A total score below 26 defines impaired sexual function.
Women's quality of sexual life evaluation - Couple Satisfaction Index-16 (CSI-16) | Preoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Couple Satisfaction Index-16 (CSI-16) questionnaire.
  CSI-16 is a precise, consistent and validated scale that evaluates the quality of a couple's relationship satisfaction. Each item is scored from 0 to 5 with different answer formats. The total score can range from 0 to 81. Higher is the total score, better is the relationship satisfaction. A relationship dissatisfaction is suggested when the total score is bellow 51,5.
Women's quality of sexual life evaluation - Couple Satisfaction Index-16 (CSI-16) | 3 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Couple Satisfaction Index-16 (CSI-16) questionnaire.
  CSI-16 is a precise, consistent and validated scale that evaluates the quality of a couple's relationship satisfaction. Each item is scored from 0 to 5 with different answer formats. The total score can range from 0 to 81. Higher is the total score, better is the relationship satisfaction. A relationship dissatisfaction is suggested when the total score is bellow 51,5.
Women's quality of sexual life evaluation - Couple Satisfaction Index-16 (CSI-16) | 6 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using the Couple Satisfaction Index-16 (CSI-16) questionnaire.
  CSI-16 is a precise, consistent and validated scale that evaluates the quality of a couple's relationship satisfaction. Each item is scored from 0 to 5 with different answer formats. The total score can range from 0 to 81. Higher is the total score, better is the relationship satisfaction. A relationship dissatisfaction is suggested when the total score is bellow 51,5.
Women's quality of sexual life evaluation - Self reported questionnaire on dyspareunia | Preoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using a self-reported questionnaire on dyspareunia.
  This questionnaire assesses presence of superficial and/or deep dyspareunia together with pain intensity. Pain intensity is assessed with the Visual Analog Scale (VAS) which rates the pain from 0 for no pain to 10 being the worst pain imaginable.
Women's quality of sexual life evaluation - Self reported questionnaire on dyspareunia | 3 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using a self-reported questionnaire on dyspareunia.
  This questionnaire assesses presence of superficial and/or deep dyspareunia together with pain intensity. Pain intensity is assessed with the Visual Analog Scale (VAS) which rates the pain from 0 for no pain to 10 being the worst pain imaginable.
Women's quality of sexual life evaluation - Self reported questionnaire on dyspareunia | 6 months postoperative
  Women's sexual Quality of Life evaluation after benigne adnexal surgery by vNOTES compared to Conventional Abdominal Laparoscopy using a self-reported questionnaire on dyspareunia.
  This questionnaire assesses presence of superficial and/or deep dyspareunia together with pain intensity. Pain intensity is assessed with the Visual Analog Scale (VAS) which rates the pain from 0 for no pain to 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Effectiveness | Peroperative
  Evaluation of the success rate (removal of the specimen without the need of conversion to laparoscopy or open-surgery) and the procedure duration including the need for adhesiolysis.
Pain evaluation | Preoperative
  Mean pain intensity will be evaluated with the Visual Analog Scale (VAS) which rates the pain intensity from 0 for no pain to 10 being the worst pain imaginable. Pain location will be assessed in a descriptive form.
Lenght of stay | During hospital stay, from day of the surgery up to 30 days after surgery
  Evaluation of lenght of stay in days ranging from 0 for the day of the intervention to 30 for the 30th day after the intervention.
Pain evaluation | During hospital stay, from day of the surgery up to 30 days after surgery
  Pain intensity will be evaluated every day with the Visual Analog Scale (VAS) which rates the pain intensity from 0 for no pain to 10 being the worst pain imaginable. Names and classes of painkillers taken will be recorded daily during hospitalisation, noting the total milligram dosage per 24 hours for each drug (class 1 for simple analgesics, class 2 for addition of morphine derivatives, class 3 for morphine and morphine derivatives).
Pain evaluation | 1 month postoperative
  Mean pain intensity will be evaluated with the Visual Analog Scale (VAS) which rates the pain intensity from 0 for no pain to 10 being the worst pain imaginable. Pain location will be assessed in a descriptive form. Assessment of analgesic intake and class of painkillers when used (class 1 for simple analgesics, class 2 for addition of morphine derivatives, class 3 for morphine and morphine derivatives).
Complications rate | Peroperative
  Failure to enter the peritoneal cavity, need for conversion, intraoperative complication during peritoneal cavity access, intraoperative blood loss, bowel or vessel injury.
Complications rate | 1 month postoperative
  Delayed vaginal or parietal healing (abscess, hematoma, dehiscence), trocar-site hernia, trocar-site nerve injury, re-hospitalization and re-operation.
Histological analysis after morcellation/aspiration of the surgical specimen | Peroperative
  Histological analysis after morcellation/aspiration of the surgical specimen : completed/ limited and diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Dubuisson, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krull E, Lambat Emery S, Viviano M, Aerts L, Petignat P, Dubuisson J. Assessment of women's sexual quality of life after benign adnexal surgery using vNOTES approach in comparison to conventional laparoscopy: protocol for a randomised controlled trial. BMJ Open. 2023 Sep 7;13(9):e073691. doi: 10.1136/bmjopen-2023-073691. PMID 37678943

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT05761275/Prot_SAP_000.pdf